CLINICAL TRIAL: NCT00187564
Title: Pilot Study on the Effect of Oral Controlled-Release Alpha-Lipoic Acid on Oxidative Stress in Adolescents With Type 1 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Stephen E. Gitelman, UCSF
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H7023-25421
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2008-05-06 (Estimated); Status verified 2005-09

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus, Type 1; lipoic acid; oxidative stress
MeSH Terms: conditions — Diabetes Mellitus, Type 1

INTERVENTIONS:
Drug: controlled-release oral alpha-lipoic acid

SUMMARY:
The long-term effects of high blood sugar include blindness, kidney failure, and nerve damage that can ultimately cause loss of limbs. Research has shown that high blood sugar increases the amount of reactive oxygen species (ROS) produced in diabetics, and that the increase in ROS causes damage to eyes, kidneys, and nerves by a process called "oxidative stress." We postulate that alpha-lipoic acid, a potent anti-oxidant, can stop ROS from forming, thereby preventing long-term complications in diabetes. In this pilot study, we will be giving 30 teenagers with type 1 diabetes (T1D) controlled-release alpha-lipoic acid for 3 months, and comparing the amount of oxidative stress before and after treatment. Ten teenagers with T1D will receive placebo instead of alpha-lipoic acid and undergo the same research protocol to aid in validation of outcome measures.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be pubertal (defined as Tanner stage II or greater), or post-pubertal, with an upper age limit of 21 years.
2. Subjects must have diabetes by 1997 ADA criteria:

   1. fasting plasma glucose >= 126 mg/dL, or
   2. 2 hour postprandial glucose >= 200 mg/dL
3. Subjects must have history of least one auto-antibody associated with T1D, either glutamic acid decarboxylase (GADA) or islet cell autoantigen 512 (ICA512), or history of diabetic ketoacidosis.

Exclusion Criteria:

1. Subjects must not have history of eye, kidney or nerve damage 2. Subjects must not be deemed unable or unlikely to comply with the protocol. Children who are unable to swallow pills, or are unwilling to take pills twice daily will be excluded from the study.

-

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40
Dates: Start 2004-08; Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
1. protein carbonyl (measurement of oxidized protein)
2. Thiobarbituric Acid Reactive Substances (TBARS) (measurement of oxidized lipid)
3. 8-Oxo-dG/8-Oxo-dA (measurement of oxidized DNA)
4. Trolox equivalent antioxidant capacity (TEAC) (measurement of total antioxidant status)

SECONDARY OUTCOMES:
1. Hb A1c
2. Urine albumin/creatinine ratio

CONTACTS AND LOCATIONS:
Overall Officials: Stephen E Gitelman, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Division of Pediatric Endocrinology, San Francisco, California, United States

REFERENCES:
- See also: UCSF Diabetes Center — http://www.diabetes.ucsf.edu/